CLINICAL TRIAL: NCT06451458
Title: ECHO for Diabetes and Multiple Chronic Conditions Study
Acronym: E4DMMC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Presbyterian Medical Services (Unknown); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Yiliang Zhu, Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-211; TE-2022C3-30560 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute)
Record Dates: First submitted 2024-05-20; First posted 2024-06-11 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus; Chronic Disease
Keywords: Diabetes; Telehealth; Hypertension; Chronic kidney disease; Hyperlipidemia; Depression; Federally Qualified Health Center (FQHC)
MeSH Terms: conditions — Diabetes Mellitus; Chronic Disease; Hypertension; Renal Insufficiency, Chronic; Hyperlipidemias; Depression

STUDY DESIGN:
Intervention Model Description: Pragmatic, Cluster Randomized Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECHO Intervention (Experimental): 10 FQHCs from the PMS health system will be randomized to the ECHO Intervention Arm. All healthcare team members in the intervention arm will attend ECHO program sessions, and the FQHCs are the primary subjects of the ECHO intervention. However, the investigators examine outcomes at both the level of the healthcare team and at the level of the patients who are empaneled to the healthcare team. Persons with DMMC cared for by the healthcare teams at the FQHC clinics are the patient population for this intervention.
  Interventions: Behavioral: ECHO program for DMMC
- Comparator (Active Comparator): 10 FQHCs from the PMS health system will be randomized to the comparator arm which is usual care. Persons with DMMC cared for by the healthcare teams at the FQHC clinics are the patient population for this comparator arm.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: ECHO program for DMMC — For the intervention, an 18-month ECHO program of weekly videoconference sessions will mentor healthcare teams on complex care strategies for patients with DMMC, emphasizing evidence-based best practices related to common chronic conditions (e.g., diabetes, CKD, hypertension, hyperlipidemia and depression). Mentorship will be provided by a multidisciplinary team of experts including a patient representative, diabetes educator, endocrinologist, psychiatrist, a nephrologist/kidney disease and hypertension specialist, a clinical pharmacist, and a cardiology consultant. Each session will consist of a didactic presentation, de-identified patient case presentations, and questions and discussion.
  Arms: ECHO Intervention
Behavioral: Usual care — The comparator will consist of 10 PMS FQHC clinics with healthcare teams practicing usual care according to PMS standard practices during the 18 months of the intervention arm.
  Arms: Comparator

SUMMARY:
Diabetes mellitus is a chronic condition that affects the body's ability to process sugar effectively, which over time can increase the risk of heart disease, high blood pressure, and kidney damage. Other chronic conditions include high cholesterol, obesity, and depression. Persons with diabetes mellitus and multiple chronic conditions (DMMC) face higher risks of losing physical or mental function, experiencing other chronic conditions, and death. Most of the residents of New Mexico (NM) belong to groups at risk for developing DMMC. Finding quality healthcare is a key factor, as NM also ranks among the largest, poorest, and most rural states. Primary care providers (PCPs) most often treat DMMC patients, but healthcare teams can lack confidence in managing these complex patients and struggle to keep up with recommended guidelines.

This Project ECHO model (ECHO) for DMMC, a telehealth intervention for healthcare teams, can lead to lower blood sugar levels in DMMC patients being treated at NM primary care clinics. ECHO is a "telementoring" program that trains healthcare teams to provide specialized medical care at their local clinics. This is done by connecting healthcare teams with specialist mentors at academic medical centers through videoconferencing sessions. During ECHO program sessions, groups of healthcare teams hear lectures on key topics in DMMC care from experts, and then give presentations of anonymous patient cases by a healthcare teams for discussion and to receive recommendations.

This clinical pragmatic trial aims to learn if the intervention will improve patient blood sugar levels in persons with DMMC who are being treated at selected health clinic sites throughout New Mexico.

The study aims to answer:

* Whether a 0.5% drop in HbA1c on average can be achieved in the group whose healthcare teams are receiving the ECHO intervention compared to the comparator group, whose providers will not receive the intervention.
* Whether the rate of an individual's HbA1c was greater than 8.5% at the baseline will be reduced by 15% at the end of the intervention.

Researchers will compare health data for patients empaneled to healthcare teams in the study and the usual care comparator group both before and after the intervention period to see whether the ECHO model has a positive influence on test results.

DETAILED DESCRIPTION:
Persons with diabetes mellitus and multiple (2+) chronic conditions (DMMC) are at increased risk of functional decline, lower quality of life, and mortality. In a state ranked among the largest, poorest, and most rural, a high proportion of the diverse residents of New Mexico (NM) belong to groups at risk for developing DMMC. Lack of access to quality healthcare is a key risk factor. Healthcare teams at Federally Qualified Health Centers (FQHCs) in medically underserved areas must have knowledge of, and be able to implement, evidence-based management guidelines to address disease complexity such as DMMC, but the healthcare teams face barriers including lack of confidence in managing complex DM and comorbid conditions and keeping up with evolving best practice guidelines. Our primary research question is whether the Project ECHO model (ECHO), a telehealth intervention for healthcare teams, can achieve significant and durable reductions in HbA1c levels relative to usual care in patients with DMMC seeking care at NM's FQHCs clinics.

Project ECHO is a "telementoring" program for remotely training healthcare teams to enable the healthcare teams to provide specialized medical care at local clinics under the ongoing mentorship of an interdisciplinary team of specialists based at academic medical centers. The ECHO model uses a combination of didactic and case-based learning to help healthcare teams, specialists, and other participants co-develop treatment plans for their patients with complex conditions. Through iterative guided practice, healthcare teams gain expertise in administering specialized medical care in primary care settings. Unlike traditional direct service or specialty consultation telehealth models, the ECHO model works on the principle of workforce multiplication, expanding access to best practice specialty healthcare by increasing healthcare team capacity to care for DMMC patients closer to their homes.

The ECHO for Diabetes and Multiple Chronic Conditions (E4DMMC) study is a cluster-randomized pragmatic trial, and will investigate the effectiveness of Project ECHO's telementoring intervention, compared to usual care practices, for optimizing the management of DMMC within vulnerable populations seeking treatment in NM FQHC clinics. E4DMMC aims to achieve, relative to the usual care arm: (1) a clinically significant ( ≥0.5%) reduction in HbA1c on average, and ≥15% reduction in rate of patients with HbA1c > 8.5% at 18-months into-intervention; (2) significant and clinically meaningful improvements on secondary clinical outcomes for other chronic conditions (blood pressure, cholesterol level, depressive symptoms, and referrals to smoking cessation); (3) similar improvements in clinical outcomes across telehealth modalities (e.g., audio-only vs. videoconference); (4) increased adoption of clinical best practices; and (5) increased patient activation and satisfaction with care. Thus, we will evaluate outcomes at both healthcare team level and at the level of patient empaneled to the healthcare team.

Our primary patient population consists of an estimated 7000 patients with DMMC actively receiving routine care from the 20 Presbyterian Medical Services (PMS) FQHC clinics with the highest patient volume and identified through PMS EHR. This population is diverse and underserved: 45% are Hispanic/Latino, and 14% are American Indian and Alaska Native; and 48% are insured through Medicaid. Across the 20 clinics, 25-48% of these patients with DM reported an HbA1c > 8.5%. Eleven clinics are in rural or mixed rural/urban counties, serving 55% of all patients with DMMC in this population. The median number of healthcare team members across these clinics is five, including clinicians, registered nurses, physician associates, and medical assistants.

The investigators will partner with PMS, the largest system of FQHC clinics in New Mexico to randomize 20 PMS FQHC clinics, 10 each to the ECHO intervention arm and Usual Care comparator arm. For the intervention, an ECHO program consisting of weekly videoconference sessions will mentor healthcare teams on complex care strategies for patients with DMMC, emphasizing evidence-based best practices related to common chronic conditions (e.g., diabetes, chronic kidney disease (CKD), hypertension, hyperlipidemia, and depression). The comparator will consist of clinical sites where healthcare teams are practicing usual care for DMMC patients, continuing standard practices for ensuring best practice care. Primary outcome data will be tracked for 21 months post-intervention in the ECHO intervention arm.

ELIGIBILITY:
Inclusion criteria:

* Twenty PMS sites with the highest patient volume.
* All members of the PMS sites (participants) healthcare teams between 18 and 89 years of age, all genders, and all ethnicities.

Exclusion criteria:

* There is no exclusion criteria.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c trajectory | At least once every 6 months per Electric Health Record (EHR), during 12 months baseline prior to intervention, during 18 months intervention.
  A decreasing trajectory in patients' HbA1c over time during and following ECHO intervention, reaching an average of 0.5% drop 18 months into intervention compared with comparator
HbA1c level in control | At least once every 6 months per Electric Health Record (EHR), during 12 months baseline prior to intervention, during 18 months intervention.
  15% decreases in per-patient rate of HbA1c>8.5% by 18 months into intervention, respectively, compared with comparator

SECONDARY OUTCOMES:
Use of any tele-med modalities for patient visits | Every encounter per EHR during 12 months baseline prior to intervention, during the study period (18 months intervention and up to 18 months follow-up for the intervention arm)
  Percentage of DMMC patients with at least 2 HbA1c tests per year as adherence to recommended DM management across modalities (audio-only vs. videoconference)
Hypertension | Per encounter; per EHR during 12 months of baseline prior to intervention, during the 18 months of intervention period and up to 18 months of follow-up
  Patient blood pressure not in control (systolic blood pressure (SBP)>130 and/or diastolic blood pressure (DBP)>80)
Cholesterol | Annual during 12 months of baseline prior to intervention, during the 18 months intervention and up to 18 months of follow-up; per EHR
  Patient low-density lipoprotein LDL-C
Kidney function | Annual during 12 months of baseline prior to intervention, during the 18 months intervention and up to 18 months of follow-up; per EHR
  Estimated glomerular filtration rate (eGFR) and/or urine albumin-creatinine ratio (UACR)
Depressive symptoms - Large version | Per encounter; per EHR during 12 months of baseline prior to intervention, during the 18 months of intervention period and up to 18 months of follow-up
  Rate of at least one positive Patient Health Questionnaire (PHQ) -2 per patient per 12-month period. The score ranges from a minimum of 0 and maximum of 6, with a higher score indicating more severe symptoms of major depressive disorder.
Depressive symptoms - Small version | Per encounter; per EHR during 12 months of baseline prior to intervention, during the 18 months of intervention period and up to 18 months of follow-up
  Depression screening score trajectory on PHQ-2 (amongst the total population and amongst those with positive PHQ-2) or PHQ-9 (only amongst those with positive PHQ-2) per 12-month period. PHQ-9 score ranges between a minimum of 0 and a maximum of 27, with the higher the score meaning a greater severity of depression.
Obesity | Per encounter; per EHR during 12 months of baseline prior to intervention, during the 18 months of intervention period and up to 18 months of follow-up
  Body mass index
Receipt of appropriate exams | Annual during 12 months of baseline prior to intervention, during the 18 months intervention and up to 18 months of follow-up; per EHR
  1. Eye exams
  2. Foot exams
Rates of prescribing DM meds in accordance with guidelines | Per encounter during 12 months baseline prior to intervention, 18 months intervention, and up to 18 months follow-up
  DM meds: metformin, sulfonylureas (glipizide, glimepiride, glyburide), glucagon-like peptide-1 receptor agonist (GLP-1RA) (patients with atherosclerotic cardiovascular disease (ASCVD)), sodium-glucose transport protein 2 inhibitors (SGLT2i) (patients with ASCVD, CKD, heart failure), thiazolidinediones (pioglitazone), GLP-1/GIP RA (tirzepatide), and insulin.
Rates of prescribing hypertension meds in accordance with guidelines | Per encounter during 12 months baseline prior to intervention, 18 months intervention, and up to 18 months follow-up
  Hypertension meds: thiazide or thiazide like diuretics, angiotensin receptor blockers (ARB), angiotensin-converting enzyme inhibitors (ACE-I), or dihydropyridine calcium channel blockers (CCB).
Rates of prescribing CKD meds in accordance with guidelines | Per encounter during 12 months baseline prior to intervention, 18 months intervention, and up to 18 months follow-up
  CKD meds: ACE-I or ARB, SGLT2i, or finerenone.
Rates of prescribing hyperlipidemia meds in accordance with guidelines | Per encounter during 12 months baseline prior to intervention, 18 months intervention, and up to 18 months follow-up
  Hyperlipidemia meds: moderate-intensity statin, OR high-intensity statin.
Rates of prescribing hypertriglyceridemia med in accordance with guidelines | Per encounter during 12 months baseline prior to intervention, 18 months intervention, and up to 18 months follow-up
  Hypertriglyceridemia meds: icosapent ethyl.
Depression care - Large and Small version | Per encounter; per EHR during 12 months of baseline prior to intervention, during the 18 months of intervention period and up to 18 months of follow-up
  Patient Health Questionnaire (PHQ) -2/PHQ-9 screening completion: PHQ-2 completion rate per primary care encounter over a 12-month period. PHQ-9 completion rate per instance of positive PHQ-2 over a 12-month period. (See Depressive Symptoms for range)
Depression care intervention | Per EHR, -12 to 0 months, 1 to 12 months, 13-24 months
  Minimally adequate treatment for depression:
  Depressive disorder diagnosis rate per patient per 12-month period.
  Amongst patients with a depressive disorder diagnosis, percentage receiving:
  two or more months of an appropriate antidepressant medication plus four or more visits to any type of prescribing provider per 12-month period, OR
  8 or more psychotherapy visits with any professional lasting an average of 30 minutes per 12-month period.
Lifestyle counseling according to guidelines | Annual during 12 months of baseline prior to intervention, during the 18 months intervention and up to 18 months of follow-up; per EHR
  1. Smoking cessation counseling
  2. Diet counseling
  3. Physical exercise counseling
Presbyterian Medical Services (PMS) Patient satisfaction survey | Per PMS standard patient survey; per encounter during 12 months of baseline prior to intervention, during 18 months of intervention and up to 18 months of follow-up
  PMS conducts routine patient satisfaction survey post each encounter. Survey is proprietary. Improvement in patient satisfaction in ECHO intervention compared with comparator. Score goes from lowest to high (scale of 1 to 5), and increase is better outcome.
Health behaviors | Per PMS standard patient survey; per encounter during 12 months of baseline prior to intervention, during 18 months of intervention and up to 18 months of follow-up
  Patient reports: (1) checking blood glucose during the last 7 days; (2) checking their feet during the last 7 days.
Tobacco use | Per PMS standard patient survey; per encounter during 12 months of baseline prior to intervention, during 18 months of intervention and up to 18 months of follow-up
  Patient reports smoking cigarettes in the last 30 days.
Diet | Per PMS standard patient survey; per encounter during 12 months of baseline prior to intervention, during 18 months of intervention and up to 18 months of follow-up
  Patient reports: (1) soda consumption in last 30 days; (2) high fat foods consumed during last 7 days; (3) spacing carbo- hydrates evenly during last 7 days
Physical exercise | Per PMS standard patient survey; per encounter during 12 months of baseline prior to intervention, during 18 months of intervention and up to 18 months of follow-up
  Patient reports physical activity of at least 30 mins during the last 7 days.

OTHER OUTCOMES:
HbA1c levels | At least once every 6 months per Electric Health Record (EHR), during 12 months baseline prior to intervention, during 18 months intervention.
  HbA1c change over intervention and follow-up for DM patients with 1 or no other chronic condition
HbA1c levels and disease progression - pre-DM | Per encounter; per EHR during 12 months of baseline prior to intervention, during the 18 months of intervention period and up to 18 months of follow-up
  HbA1c change over intervention and follow-up for pre-DM patients
HbA1c levels and disease progression - newly diagnosed DM | At least once every 6 months per Electric Health Record (EHR), during 12 months baseline prior to intervention, during 18 months intervention.
  HbA1c change over intervention and follow-up for newly diagnosed DM or DMMC patients who did not have baseline data
Patient Activation Measure (PAM) | Per PMS standard patient survey; during 12 months of baseline prior to intervention, during 18 months of intervention and up to 18 months of follow-up
  Short form 13-item Patient Activation Measure. The scale is proprietary, and there is no low or high.

CONTACTS AND LOCATIONS:
Overall Officials: Yiliang Zhu, PhD, Principal Investigator — University of New Mexico Health Science Center; Matthew Bouchonville, MD, Principal Investigator — University of New Mexico Health Science Center; Vallabh Shah, PhD, Study Director — University of New Mexico Health Science Center
Locations (1):
- Presbyterian Medical Services, Santa Fe, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
We will follow PCORI's Policy for Data Management and Data Sharing.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Callis PD, Santini A. A suggested role for polymorphonuclear leukocytes in the perpetuation of periapical disease. Oral Surg Oral Med Oral Pathol. 1985 Jan;59(1):88-90. doi: 10.1016/0030-4220(85)90122-7. PMID 3856208
- [Background] Arora S, Kalishman SG, Thornton KA, Komaromy MS, Katzman JG, Struminger BB, Rayburn WF, Bradford AM. Project ECHO: A Telementoring Network Model for Continuing Professional Development. J Contin Educ Health Prof. 2017 Fall;37(4):239-244. doi: 10.1097/CEH.0000000000000172. PMID 29189491
- [Background] Arora S, Thornton K, Murata G, Deming P, Kalishman S, Dion D, Parish B, Burke T, Pak W, Dunkelberg J, Kistin M, Brown J, Jenkusky S, Komaromy M, Qualls C. Outcomes of treatment for hepatitis C virus infection by primary care providers. N Engl J Med. 2011 Jun 9;364(23):2199-207. doi: 10.1056/NEJMoa1009370. Epub 2011 Jun 1. PMID 21631316
- [Background] MATTHEW F. BOUCHONVILLE, ERIK B. ERHARDT, YURIDIA L. LEYVA, LARISSA MYASKOVSKY, MARK L. UNRUH, SANJEEV ARORA; 1029-P: Building Diabetes Care Capacity in Rural Underserved Communities-A Comparison of Cardiorenal Risk Factor Outcomes in Patients Treated by ECHO-Trained Providers vs. an Academic Medical Center. Diabetes 20 June 2023; 72 (Supplement_1): 1029-P. https://doi.org/10.2337/db23-1029-P
- [Background] Bouchonville MF, Hager BW, Kirk JB, Qualls CR, Arora S. ENDO ECHO IMPROVES PRIMARY CARE PROVIDER AND COMMUNITY HEALTH WORKER SELF-EFFICACY IN COMPLEX DIABETES MANAGEMENT IN MEDICALLY UNDERSERVED COMMUNITIES. Endocr Pract. 2018 Jan;24(1):40-46. doi: 10.4158/EP-2017-0079. PMID 29368967
- [Background] Bouchonville MF, Paul MM, Billings J, Kirk JB, Arora S. Taking Telemedicine to the Next Level in Diabetes Population Management: a Review of the Endo ECHO Model. Curr Diab Rep. 2016 Oct;16(10):96. doi: 10.1007/s11892-016-0784-9. PMID 27549110
- [Background] Nelson RG, Pankratz VS, Ghahate DM, Bobelu J, Faber T, Shah VO. Home-Based Kidney Care, Patient Activation, and Risk Factors for CKD Progression in Zuni Indians: A Randomized, Controlled Clinical Trial. Clin J Am Soc Nephrol. 2018 Dec 7;13(12):1801-1809. doi: 10.2215/CJN.06910618. Epub 2018 Nov 15. PMID 30442864
- [Background] Paul M, Davila Saad A, Billings J, Blecker S, Bouchonville MF, Berry C. MON-190 Endo ECHO Improves Patient-Reported Measures of Access to Care, Health Care Quality, Self-Care Behaviors, and Overall Quality of Life for Patients with Complex Diabetes in Medically Underserved Areas of New Mexico. J Endocr Soc. 2019 Apr 30;3(Suppl 1):MON-190. doi: 10.1210/js.2019-MON-190. PMCID: PMC6551170.